CLINICAL TRIAL: NCT04706988
Title: Relationship of Airway Microbiota, Endotype and Phenotype in Adult Asthma
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Honorary Associate Professor, Chinese University of Hong Kong
Other Study IDs: Asthma microbiome_v01
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal flock swab of asthma subjects. The swabs will be subjected to sequence analysis of 16S rRNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Treatment of asthma according to GINA guideline — Pharmacological treatment depending on level of control of asthma

SUMMARY:
Increasing evidence supports that the respiratory microbiota, including viral and bacterial microorganisms, play important roles in respiratory health and disease. Microbial patterns in airways may induce distinctive endotypes of asthma. Previous studies suggest host-microbiota interactions in children may account for the heterogeneity of endotypes and clinical presentations. However, information on such relationship is limited in adults. Furthermore, how the upper airway microbiome is related to asthma endotype and phenotype is not well understood. Knowledge of microbiota in the airway allows exploration of therapeutic manipulation of the microbiome and targeting the development of asthma prevention strategies and the optimization of asthma treatment.

DETAILED DESCRIPTION:
This study plans to assess microbes in nasopharyngeal flock swab of asthma subjects. The swabs will be subjected to sequence analysis of 16S rRNA. Endotypes (e.g. TH1 vs TH2 inflammation) and phenotypes of the subjects (e.g. severity, exacerbation, lung function, etc.) will be assessed. The planned sample size is 140 adult asthma subjects. Patients will have nasopharyngeal swabs taken at baseline, 3 months (after optimization of asthma treatment at baseline) and at 1 year. They will undergo assessments, including clinical course, lung function, exhaled nitric oxide, skin test, and blood test (including eosinophils and immunoglobulin E levels). All subjects will be followed up for 2 years to assess subsequent exacerbations and levels of asthma control. The 16S data retrieved from the official website of HMP (http://www.hmpdacc.org/) will be used as the geographic reference for this study. Sequences assigned to different taxonomic levels, from phylum to genus using the RDP (ribosomal database project) database, will be clustered into operating taxonomic units (OTUs). Bioinformatic tools will be used to assess the relations of microbiota, asthma endotypes and phenotypes and change of microbiota pattern upon optimization of asthma drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 80 years and have a diagnosis of asthma according to the Global Initiative for Asthma (GINA) document in 2020.
* Asthma is defined as those with a consistent history and prior documented evidence of variable airflow obstruction, with evidence of an increase in FEV1 greater than 12% or 200 mL following bronchodilator or bronchial hyperresponsiveness on bronchial provocation testing, when stable.

Exclusion Criteria:

* Patients with respiratory diseases with other known respiratory diseases including chronic obstructive pulmonary disease, bronchiectasis, tuberculosis (TB)-destroyed lung parenchyma, history of lung resection and lung cancer
* Individuals older than 40 years with a smoking history of more than 10 pack-years or significant biomass exposure
* Patients currently randomized in other clinical studies
* Pregnant women
* Current smokers (who have not quit smoking in the past 1 year)
* Systemic and intranasal antibiotics treatment within 4 weeks
* Signs and symptoms of respiratory tract infections (upper or lower) within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma subjects
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome pattern | 12 months
  The 16S data retrieved from the official website of HMP (http://www.hmpdacc.org/) will be used as the geographic reference for this study. Sequences assigned to different taxonomic levels, from phylum to genus using the RDP database, will be clustered into operating taxonomic units (OTUs) based on their best BLAST hit to reference type strain 16S DNAs at 98% sequence identity cutoff.

SECONDARY OUTCOMES:
disease severity | 12 months
  GINA treatment steps
Asthma control | 12 months
  Level of asthma control
Lung function | 12 months
  FEV1 % predicted
endotype (eosinophilic vs neutrophilic asthma) | 12 months
  Blood eosinophil and IgE level

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Ko, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No